CLINICAL TRIAL: NCT06072014
Title: Developing Immersive Gamification Technology Systems for the Management of Patients With Alzheimer's Disease With Behavioral and Psychological Symptoms of Dementia (Phase 2 Trial)
Brief Title: ImGTS for Patients With Behavioral and Psychological Symptoms of Dementia (Phase 2)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Augmented eXperience E-health Laboratory (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AXEL0003
Record Dates: First submitted 2023-09-28; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Dementia Alzheimers
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Head-mounted display (HMD) (Experimental): The HMD system uses a commercially available virtual headset, the Oculus/Meta Quest 2, which allows a user to view a virtual environment in 360 degrees and to interact with the environment using hand-tracking technology (i.e., when a user's hand is projected into the virtual world to be used for interactions and gestures).
  Interventions: Other: Virtual reality
- Semi-cave automatic virtual environment (semi-CAVE) (Experimental): The semi-CAVE system uses projectors and projector screens to provide a 270-degree view of the virtual environment. These projectors are connected to a powerful workstation (desktop computer), which uses HTC Vive trackers and base stations to track user movements and interactions
  Interventions: Other: Virtual reality

INTERVENTIONS:
Other: Virtual reality — A role-playing game with activities based on existing therapy activities (such as orientation therapy, reminiscence therapy, art therapy, and music therapy) that are used to manage behavioral and psychological symptoms of dementia

SUMMARY:
The proposed research project aims to answer the question "Are immersive technology systems effective in the management and treatment of patients with BPSD?". This project is composed of three phases and the current study is the second phase. The phase 2 trial aims to create an immersive technology system for managing the behavioral and psychological symptoms of dementia and determine its clinical effectiveness, safety, usability, and acceptability among patients with mild to moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years old or older
* Diagnosed with mild to moderate Alzheimer's dementia according to the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria
* Montreal Cognitive Assessment-Philippines (MOCA-P) score of 10-20 inclusive
* Neuropsychiatric Inventory (NPI-12) score 1-50 inclusive
* Reisberg Scale Stage 4-5 inclusive
* Stable dose of antidepressants for the past 6 weeks
* Stable dose of antipsychotics for the past 4 weeks
* Able to walk unassisted or with minimal assistance, with or without assistive device
* No other explanation for condition based on reasonable clinical diagnostics

Exclusion Criteria:

* Have mild cognitive impairment (no dementia)
* Have MOCA-P score less than 10 or more than 20
* Other non-amnestic dementia syndromes
* Have receptive aphasia
* Have significant visual or hearing impairment
* Have an active psychiatric disorder prior to Alzheimer dementia diagnosis
* Had previous episodes of seizures, diagnosis of epilepsy, or intake of antiepileptic or seizure medications
* Have quadriplegia or paralysis of the dominant hand
* Have a history of motion sickness
* Experience claustrophobia
* Have a diagnosis of a terminal illness or a life expectancy of less than one year

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of behavioral and psychological symptoms of dementia will be assessed using the Neuropsychiatric Inventory-12 | Within one hour after completion of the fourth session
  The NPI evaluates the degree and severity of BPSDs and the distress it causes the primary caregiver. Scores range from 0 to 120 where higher scores indicate greater psychiatric disturbance.
Incidence of virtual reality sickness symptoms will be assessed using the Virtual Reality Sickness Questionnaire | Immediately after each intervention, within an hour of completion of the virtual reality game
  The VRSQ will measure a participant's experience with the following symptoms: general discomfort, fatigue, eye strain, difficulty focusing, headache, fullness of head, blurring of vision, dizziness (when eyes are closed), and vertigo. Symptoms will be rated on a 4-point scale: 0 or None, 1 or Slight, 2 or Moderate, and 3 or Severe.
Usability of the virtual reality intervention will be assessed using the System Usability Scale | Immediately after each intervention, within an hour of completion of the virtual reality game
  The SUS is a 10-item questionnaire that is widely used in the evaluation of various kinds and aspects of technology. Each question has five response options ranging from 'Strongly agree' to 'Strongly disagree', which has a corresponding number value. Each response is added and multiplied by 2.5 to obtain the final score that ranges from 0 to 100. A SUS score above 68 is considered above average.

SECONDARY OUTCOMES:
Cognitive function will be assessed using MOCA-P | Within one hour after completion of the fourth session
  Montreal Cognitive Assessment-Philippines (MOCA-P) is a 30-item test that takes about 10-12 minutes to complete. The test measures different cognitive domains such as visuospatial/executive, naming, memory, attention, language, abstraction, and orientation.
Cognitive function will be assessed using MMSE | Within one hour after completion of the fourth session
  The Mini-Mental State Exam (MMSE) is a 30-item test for cognitive function. It assesses attention, orientation, memory, registration, recall, calculation, language, and an individual's ability to draw a complex polygon.
Cognitive function will be assessed using ADAS-Cog | Within one hour after completion of the fourth session
  The cognitive subscale of the Alzheimer's Disease Assessment Scale (ADAS-Cog) is an 11-item tool for the assessment of the following tasks: word recall, naming objects and fingers, commands, constructional praxis, ideational praxis, orientation, word recognition, and language.
Activities of daily living will be assessed using ADCS-ADL | Within one hour after completion of the fourth session
  The Alzheimer's Disease Cooperative Study - Activities of Daily Living Inventory (ADCS-ADL) is a 24-item assessment on activities of daily living within the past four weeks
Health-related quality of life will be assessed using DEMQOL | Within one hour after completion of the fourth session
  The Health-related quality of life for people with dementia (DEMQOL) is a 28-item self-report measure of quality of life specific for persons with mild-to-moderate dementia. It covers four dimensions of quality of life, namely, daily activities, memory, negative emotion, and positive emotion.

OTHER OUTCOMES:
Acceptability | Within one day after completing virtual reality experience
  Acceptability will be measured among a small group of patients and their caregivers through an interview and a focus group discussion

CONTACTS AND LOCATIONS:
Overall Officials: Veeda Michelle M. Anlacan, MD, Principal Investigator — University of the Philippines Manila
Locations (1):
- University of the Philippines College of Allied Medical Professions Immersive Technology Laboratory, Manila, National Capital Region, Philippines

REFERENCES:
- [Background] Anlacan, V.M.M. et al. (2023). Application Design for a Virtual Reality Therapy Game for Patients with Behavioral and Psychological Symptoms of Dementia. In: Krouska, A., Troussas, C., Caro, J. (eds) Novel & Intelligent Digital Systems: Proceedings of the 2nd International Conference (NiDS 2022). NiDS 2022. Lecture Notes in Networks and Systems, vol 556. Springer, Cham. https://doi.org/10.1007/978-3-031-17601-2_15